CLINICAL TRIAL: NCT00231348
Title: Nefazodone in the Treatment of Social Phobia: Functional Brain Imaging and Neuroendocrine Correlates
Brief Title: Nefazodone in the Treatment of Social Phobia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0707-1997
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Social Anxiety Disorder (SAD)
Keywords: Social anxiety disorder; social phobia; positron emission tomography (PET; regional cerebral blood flow (rCBF); nefazodone; amygdala
MeSH Terms: conditions — Phobia, Social | interventions — nefazodone

INTERVENTIONS:
Drug: Nefazodone

SUMMARY:
The purpose of this study is to determine the effectiveness of nefazadone in patients with social anxiety disorder (SAD).

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy of the 5HT2 receptor antagonist nefazadone in SAD, and to explore regional cerebral blood flow in patients with SAD when confronted with a personal phobic stimulus, using positron emission tomography (PET). Changes in cerebral blood flow were correlated with self-rated anxiety measures.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of generalized social anxiety disorder, males and females between the ages of 18-65

Exclusion Criteria:

* A history of bipolar disorder, psychotic illness, or any other anxiety disorders, organic brain disease or active drug or alcohol abuse within one year as assessed by the SCID-P and interview, or a concurrent medical condition that would not be compatible with the study in the opinion of the principal investigator. Patients required to be free of psychotropic or beta-blocker medication for 2 weeks prior to study. Pts taking fluoxetine required to be drug-free for 6 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Nemeroff, MD, PhD, Principal Investigator — Emory University Department of Psychiatry and Behavioral Sciences; Clinton D Kilts, PhD, Study Director — Emory University Department of Psychiatry and Behavioral Sciences; Jeffrey Newport, MD, Study Director — Emory University Department of Psychiatry and Behavioral Sciences
Locations (1):
- Emory University Depatment of Psychiatry and Behavioral Sciences, Atlanta, Georgia, United States